CLINICAL TRIAL: NCT01990417
Title: Evaluation of Passive Stretching in the Hamstrings Flexibility of Who Practice Exercises
Brief Title: Evaluation of Passive Stretching in the Hamstrings Flexibility
Acronym: EPSHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fortaleza University (Other)
Responsible Party: Principal Investigator, Ana Paula de Vasconcellos Abdon, PhD, Fortaleza University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: EPS-1310
Record Dates: First submitted 2013-10-13; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Students; Healthy Volunteers
Keywords: Muscle Stretching Exercises; Joint range of motion; Resistance Training; Physical Therapy
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Passive stretching (Experimental): After evaluation, the participants were randomly divided into four groups: A, B, C and D. Group A. stretched before and after workout ; group B stretched only before workout; group C stretched only after workout; and group D did not stretch at all.
  Interventions: Other: Passive stretching

INTERVENTIONS:
Other: Passive stretching — Passive stretching of the hamstrings was performed only once, lasting 30 seconds, and initiated on the right leg. Participants were in supine position with head, trunk and arms aligned along the body. The researcher remained ipsilateral to the subject´s leg being stretched and applied external force to the limit tolerated by the participant. The researcher performed a hip flexion, knee extension, and dorsiflexion of the ankle while the opposite leg remained extended on the ground.

SUMMARY:
The present study aimed to analyze the influence of passive stretching before and after strength training on flexibility of the hamstrings in people who work out

DETAILED DESCRIPTION:
Question: Does passive stretching before and after strength training effect the flexibility of the hamstrings in people who work out?

Design: Intervention study in humans

Participants: 40 healthy student volunteers, ranging in age from 18 to 35 years old, who work out.

Intervention: The Wells bench was used to assess the flexibility of the hamstring muscle. In this test, a person sits on a mat, with the soles of both feet maintaining contact with a box. The top of the box has an indicator marked in centimeters that is used to measure flexibility by how far the person can push the indicator without bending the legs. The knees of the seated person are extended while the hips are flexed. The subject is then asked to take a deep breath, and during exhalation, flex the trunk forward with the upper limbs extended.

The upper limbs are supported by a bench of 23 cm long aligned with a tape measure over the bench. During flexion of the trunk, the right hand is placed over the left and the tips of the fingers touch the indicator on top, and move it forward as far as possible.

ELIGIBILITY:
Inclusion Criteria:

* The healthy students volunteers who worked out at the gym between 1-15 months of activities and ranging in age from 18 to 35 years

Exclusion Criteria:

* Volunteers who had history of chronic disease diagnosed and /or musculoskeletal injury.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2010-12; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
hamstrings flexibility | 30 seconds of maintenance
  After evaluation, the participants were randomly divided into four groups: A, B, C and D. Group A. stretched before and after workout ; group B stretched only before workout; group C stretched only after workout; and group D did not stretch at all.
  Passive stretching of the hamstrings was performed only once, lasting 30 seconds, and initiated on the right leg. Participants were in supine position with head, trunk and arms aligned along the body. The researcher remained ipsilateral to the subject´s leg being stretched and applied external force to the limit tolerated by the participant. The researcher performed a hip flexion, knee extension, and dorsiflexion of the ankle while the opposite leg remained extended on the ground.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Paula V Abdon, PhD, Study Director — University of Fortaleza - UNIFOR
Locations (1):
- Núcleo de Atenção Médica Integrada (NAMI), in the evaluation room of the academy school at the University of Fortaleza (UNIFOR), Fortaleza, Ceará, Brazil